CLINICAL TRIAL: NCT03638908
Title: A Phase 2, Open-label, Clinical Trial of Fluoxetine, a Selective Serotonin Reuptake Inhibitor, in the Treatment of Pulmonary Arterial Hypertension
Brief Title: Fluoxetine in Pulmonary Arterial Hypertension (PAH) Trial
Acronym: PAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIKK23; STU 082013-045 (Other: UTSouthwestern Medical Center)
Record Dates: First submitted 2018-07-12; First posted 2018-08-20 (Actual); Results first posted 2019-10-07 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluoxetine (Other): Dosing will be
  * Week 1-4: 20 mg daily
  * Week 5-8: 40 mg daily
  * Week 9-12: 60 mg daily
  * Week 13-24: 80 mg daily
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine

SUMMARY:
This protocol describes an open-label phase 2 clinical trial of fluoxetine in PAH looking at change in pulmonary vascular resistance (PVR) as the primary endpoint.

In this open-label clinical trial, 18 patients with pulmonary arterial hypertension will be given fluoxetine for 24 weeks. A Right Heart Catheterization will be performed at baseline and 24 weeks. Change in PVR will be the primary endpoint; other hemodynamic endpoints, quality of life, QIDS-SR depression scale, functional class and six-minute walk distance will also be evaluated.

Primary Hypothesis: Fluoxetine treatment for 24 weeks will lead to significantly lower pulmonary vascular resistance in 18 patients with PAH in patients treated in an open-label clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. WHO Group I PAH subtypes of idiopathic PAH and PAH associated with drugs / toxins, connective tissue disease, repaired congenital heart disease and unrepaired atrial septal defect
2. Age 16-80
3. WHO Functional Class II or III
4. Right Heart Catheterization within 3 weeks of study entry with mPAP ≥ 25 mmHg, wedge ≤ 15 mmHg, and PVR ≥ 3 Wood units.
5. Contraception use, (-) urine pregnancy test, not breast feeding (women of childbearing potential)
6. One or more approved PAH therapies for ≥ 3 months, no change in dose for 1 month (endothelin-1 antagonist, phosphodiesterase-5 inhibitor, prostacyclin / prostacyclin analog). Novel approved therapies in one of the three existing classes will also be acceptable as background therapy if they become available during the course of the study; other medication classes are excluded

   Exclusion Criteria:
7. WHO Functional Class IV or listed for lung transplant
8. Moderate or greater obstructive lung disease: FEV1/FVC <70% and FEV1 <60%
9. Moderate or greater restrictive lung disease: TLC or FVC <60% (if 50-60%: OK if TLC or FVC ≥50% + PFT stable x1 year + CT with no more than mild lung disease)
10. Other cause for pulmonary hypertension: all other WHO group I diseases (including but not limited to liver disease, HIV), and WHO Groups II-V (i.e. left heart disease, lung disease, chronic PE and miscellaneous causes)24.

    1. High probability VQ or positive CTA
    2. Left ventricular ejection fraction <40%
11. Depression
12. Severe liver, renal or other medical or physical disease preventing completion of the study procedures
13. Use of antidepressants within 3 months

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-11; Primary Completion 2017-05 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Chin, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited solely from the clinic from November 2013 to November 2016
Pre-assignment Details: This was an open label study and all subjects were assigned to receive Fluoxetine.
Groups:
- Fluoxetine: Dosing will be
  * Week 1-4: 20 mg daily
  * Week 5-8: 40 mg daily
  * Week 9-12: 60 mg daily
  * Week 13-24: 80 mg daily
  Fluoxetine
Period: Overall Study
Arm/Group | Fluoxetine
Started | 8
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fluoxetine
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: White non-hispanic | 5
  Race/ethnicity: Hispanic | 3
  Race/ethnicity: African American | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Vascular Resistance (PVR)
Description: Change in PVR between baseline and follow-up will be utilized. PVR is calculated as [(Pulmonary Artery mean - wedge) / Fick Cardiac Output]. Fick CO will be used in computing PVR over thermodilution because Fick appears to have greater precision (but not accuracy). The calculation of PVR above is measured in woods unit. Change is derived by getting the difference between baseline and week 24 PVR (Week 24 minus Baseline). mean is then computed by getting the average of the change
Time Frame: Baseline and Week 24
Population: 6 out of the 8 subjects enrolled had complete- baseline and week 24- data for analysis
Measure: Mean (Standard Deviation); unit: woods unit
Arm/Group | Fluoxetine
Number analyzed (Participants) | 6
woods unit | 6.7 (2.7)

2. Secondary Outcome: 5-HIAA (HYDROXYINDOLE ACETIC ACID) Level
Description: Urine for spot urine 5-HIAA will be collected at baseline and Week 24. Subjects will be on diet restriction 72 hours prior to urine collection. Sample will be the first morning urine on the visit day. Sample will be brought to site and then sent to affiliate outside laboratory for processing. 5HIAA results are expressed as a ratio to creatinine excretion in the unit "mg/g creatinine" Change 5-HIAA is derived by getting the difference between baseline and week 24 5HIAA results (Week 24 minus Baseline). mean is then computed by getting the average of the change
Time Frame: Baseline and Week 24
Population: unable to adequately analyze outcome as there were several missing data- values provided below are not meaningful.
Measure: Mean (Standard Deviation); unit: mg/g CRT
Arm/Group | Fluoxetine
Number analyzed (Participants) | 5
mg/g CRT | 0.375 (0.182)

3. Other Pre Specified Outcome: Markers of Platelets and Endothelial Activation in PAH.
Description: About 20ml blood will be obtained for plasma and serum at Baseline and Week 24. This will be placed in a red-top tube (serum, at least 1 ml) and blue-top tube. For the plasma tests, a plasma volume of 750 microL is required. Samples will be sent together, as a batch of 50 is required, on dry ice via overnight courier. Plasma will be obtained by drawing blood into a blue-top citrated tube, inverting the tube 6 times, and then centrifuging at 2000g for 10 minutes. The platelet poor plasma will be drawn off, and then re-centrifuged for 10 minutes before freezing.
Time Frame: Baseline and Week 24
Population: unable to analyze outcome as this sub-study was dependent on obtaining additional funding- samples were collected but not processed to provide result
Groups:
- Fluoxetine- Baseline: Dosing will be
  * Week 1-4: 20 mg daily
  * Week 5-8: 40 mg daily
  * Week 9-12: 60 mg daily
  * Week 13-24: 80 mg daily
Arm/Group | Fluoxetine- Baseline
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Exercise Capacity
Description: Exercise capacity will be measure using the 6-minute walk test. Data collected at baseline and 24 were analyzed. The test will follow the ATS guidelines for 6MWT at all time.
Time Frame: baseline and 24
Population: 6 out of total enrolled had complete data for analysis
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Fluoxetine- Baseline: subject data at baseline
- Fluoxetine- Week 24: subject data at week 24
Arm/Group | Fluoxetine- Baseline | Fluoxetine- Week 24
Number analyzed (Participants) | 6 | 6
meters | 380 (80.7) | 393 (78.6)

5. Other Pre Specified Outcome: Functional Class
Description: Functional class will be measured using the WHO functional class assessment. This is graded from WHO FC I to FC IV. Assessment will be completed by an investigator on the study at every visit.
Time Frame: baseline and 24
Population: analysis was not done as study primary endpoint was not met- since primary endpoint was not met, no further analyses were completed
Arm/Group | Fluoxetine
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Quick Inventory of Depressive Symptomatology
Description: Patient reported outcome will be assessed using the Quick Inventory of Depressive Symptomatology (16-Item) (Self-Report) (QIDS-SR16) completed at baseline, week 12 and Week 24; baseline and week 24 reported. Each question is scored from minimum of 0 to a maximum of 3; total score ranges from 0 to 42. With zero being better outcome and 42 being severe outcome
Time Frame: baseline and Week 24.
Population: 7 subjects of the total enrolled were included in the descriptive analysis. 1 subject did not complete the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fluoxetine- Baseline | Fluoxetine- Week 24
Number analyzed (Participants) | 7 | 7
score on a scale | 4.7 (2.3) | 4.3 (3.3)

7. Other Pre Specified Outcome: Patient Global Impression of Severity - Symptoms (PGIS)
Description: PGIS questionnaire will be administered for global assessment of severity. This questionnaire is categorical and measures outcome from "none" being best outcome to "severe" being the worst outcome
Time Frame: baseline
Population: as for outcome 5
Arm/Group | Fluoxetine
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Clinician Global Impression of Severity - Symptoms (CGIS)
Description: Global assessment of severity will be determined using Clinician global impression of severity - symptoms (CGIS). This questionnaire is categorical and measures outcome from "none" being best outcome to "severe" being the worst outcome
Time Frame: Week 12 and Week 24.
Population: as for outcome 5
Arm/Group | Fluoxetine
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Short Form 36
Description: Patient reported outcome will also be assessed using SF-36 completed at baseline, Week 12 and Week 24. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health
Time Frame: baseline, Week 12 and Week 24.
Population: as for outcome 5
Arm/Group | Fluoxetine
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Clinician Global Impression of Change (CGI-change)
Description: CGI-change questionnaire will be completed for global assessment of severity. This questionnaire is categorical and measures outcome from "very much better" being best outcome to "very much worse" being the worst outcome
Time Frame: Weeks 12 and 24
Population: as for outcome 5
Arm/Group | Fluoxetine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Fluoxetine
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluoxetine (N=8)
headaches (General disorders) | 4
excessive yawning (General disorders) | 2
anxiety (Psychiatric disorders) | 2
diarrhea (Gastrointestinal disorders) | 3
acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 2
fatigue (General disorders) | 2
increased palpitations (Cardiac disorders) | 2
dizziness (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT03638908/Prot_SAP_000.pdf